CLINICAL TRIAL: NCT04572321
Title: Youth Depression and Suicide Research Network
Acronym: YDSRN
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2020-0665
Record Dates: First submitted 2020-09-17; First posted 2020-10-01 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Depression; Suicide; Suicidal Ideation; Suicide, Attempted; Depressive Disorder; Depressive Symptoms; Depressive Episode; Depression and Suicide; Depression, Teen; Depression, Anxiety
Keywords: depression; suicide; suicidal ideation; suicide attempt; teen; child; depressive episode; depression in teens
MeSH Terms: conditions — Depression; Suicide; Suicidal Ideation; Suicide, Attempted; Depressive Disorder; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to build the Texas Youth Depression and Suicide Research Network to support the development of a Network Participant Registry and characterization of systems and interventions to examine statewide population health outcomes. All 12-13 sites represented in the Texas Child Mental Health Care Consortium (https://www.utsystem.edu/pophealth/tcmhcc/) have been invited to participate in the Texas Youth Depression and Suicide Research Network as "Nodes." 12 Nodes have been selected for this project. Each Node has obtained support of senior institutional leadership including the department chair. Leadership from each Node provided input and edits in the study design process by committee, with a focus on the inclusion of the "end user" in design decisions. Nodes will work closely with the Network Hub leadership to recruit, monitor, and retain participants. This will require active engagement and sustained relationships with clinics within the academic medical center as well as clinics in the community (i.e., psychiatry, psychology, counselling).

DETAILED DESCRIPTION:
Objective: To build the Texas Youth Depression and Suicide Research Network to support the development of a Network Participant Registry and characterization of systems and interventions to examine statewide population health outcomes.

Methodology: Youth patients of participating clinics (ages 8-20) and their parents will be recruited for participation in the Network Participant Registry Study. Upon informed consent/assent, baseline data will be collected regarding mood symptoms, suicidal ideation and behavior, associated comorbidities, treatment history, services use, and social determinants of health. Youth participants and parents will be sent monthly measures through the Electronic Data Capture (EDC) system developed and maintained by UT Southwestern. Additionally, measures will be given at provider visits to support delivery of measurement-based care within the clinics.

Number of Participants: 5000 Participants and/or Coupled Participants (coupled-Parent and Youth)

Criteria for Inclusion: This study will enroll youth with depression and/or suicidal ideation. and meet all of the following criteria:

* Be 8 to 20 years of age at the time of enrollment;
* Have a positive screen for depression (e.g., based on PHQ-2 (score ≥3) and/or PHQ-A of 10 or greater, OR positive for suicidal ideation or behavior (e.g., based on CHRT-SR or PHQ-A item 9); OR be in treatment for depression;
* Be willing to provide consent/assent (parents/LAR or young adult participant, aged 18-20, must be willing to provide consent; youth, aged 8-17, must be willing to provide assent);
* Be able to read, write and speak English or Spanish sufficiently to understand the study procedures and provide written informed consent to participate in the study;
* Be willing to dedicate appropriate time to complete scheduled study assessments and measures (both parent/LAR and youth).
* Be able to provide a reliable means of contact.

Visit Schedule: Screening, Baseline, 13 Follow-Up Visits (5 assessment visits with self-reports, and 8 self-report visits only) during the first two years. Four Follow-Up Visits each year in Year 3 through Year 10 (1 assessment visit with self-report and 3 self-report visits only). All visits may be conducted remotely or in person.

Outcome Measures: Multiple streams of outcome measures will be utilized for this protocol, including self-report and parent-report measures, research assessor-completed measures, clinic level measures, and data obtained through chart review from the EHR.

Safety and Tolerability Measures: Adverse event (AE) recording, 9 item Patient Health Questionnaire (PHQ-A), Concise Health Risk Tracking Self Report (CHRT)-SR.

Statistical Justification: The goals of the statistical analyses includes the following:

* To provide a descriptive summary of the data by participating network nodes as well as by various socio-demographic characteristics of the participants such as age groups, sex, urban or rural, degree of fidelity to MBC, etc.
* To build predictive models for treatment outcomes and trajectories of disease course as well as models to assist with treatment selection that may benefit subgroups of participants.

ELIGIBILITY:
Inclusion Criteria:

1. Be 8 to 20 years of age;
2. Have a positive screen for depression (e.g., based on PHQ-2 (score ≥3) and/or PHQ-A of 10 or greater, OR positive for suicidal ideation or behavior (e.g., based on CHRT-SR or PHQ-A item 9); OR be in treatment for depression;
3. Be willing to provide consent/assent (parents/LAR/guardian or young adult participant, aged 18-20, must be willing to provide consent; youth, aged 8-17, must be willing to provide assent);
4. Be able to read, write and speak English or Spanish sufficiently to understand the study procedures and provide written informed consent to participate in the study;
5. Be willing to dedicate appropriate time to complete scheduled study assessments and measures (both parent/LAR/guardian and youth).
6. Be able to provide a reliable means of contact.

Exclusion Criteria:

1. Have an acute medical or psychological condition(s) that that would, in the judgment of the study medical clinician, make participation difficult or unsafe;
2. Have an acute medical or psychological condition(s) that would result in an inability to accurately complete study requirements (e.g., neurological conditions or significant neurodevelopmental concerns);
3. Have active psychotic symptoms resulting in altered mental status and inability to provide assent or requiring immediate attention and/or higher level of intervention;
4. Have a parent/LAR/guardian who is deemed cognitively unable to provide consent (if youth participant, aged 8-17).

Ages: 8 Years to 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Participants between the ages of 8 - 20 year-olds who either have symptoms of depression, or have suicidal ideation and/or behavior, or are in treatment for depression.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2032-08 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Network participant registry | 10 years
  A participant registry with population health outcomes for youth with depression and or suicidal ideation or behavior.

SECONDARY OUTCOMES:
Predictive models | 10 years
  Develop predictive models for short and long term outcomes for youth with depression and or suicidal behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Trivedi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States